CLINICAL TRIAL: NCT02585349
Title: Cognition and Affect After Stroke: a Prospective Evaluation of Risks
Acronym: CASPER
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 12-3-068
Record Dates: First submitted 2014-12-11; First posted 2015-10-23 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Vascular Cognitive Impairment; Post-stroke Depression; Post-stroke Apathy; Post-stroke Dementia; Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Buffycoats from EDTA tubes are taken for DNA extraction (ApoE, CLU, PICALM, CR1, ACE, MTHFR). One PAXgene tube is collected to ensure long-term stability of RNA. Extraction of RNA and subsequent analysis of expression of inflammatory and stroke-related genes at the mRNA level will be done.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First-ever and recurrent ischemic and hemorrhagic stroke: First-ever and recurrent ischemic and hemorrhagic stroke patients are enrolled in the study. Recurrent strokes are only included if the patient is fully recovered from the previous event, which occurred at least 3 years ago, without obvious residual symptoms.

SUMMARY:
Stroke is a leading cause of disability, affecting about 34,000 to 41,000 individuals in the Netherlands of middle and old age every year. Due to the aging of the population, this figure will increase considerably over the next decades (Struijs et al., 2005). Twenty-five percent of stroke patients die within one month, making stroke a major risk factor for premature death in developed countries. According to the World Health Organization, stroke is the third leading cause of the burden of disease in middle and high-income countries (World Health Organization, 2008). It has a significant negative impact on quality of life of both the patients as well as their caregivers and significant others. Surviving stroke patients often struggle with its manifold and lifelong lasting consequences, with 35 percent of patients being functionally dependent one year after stroke (Wolfe, 2000) and cognitive and emotional changes which are found up to two years post-stroke (Rasquin, Lodder, & Verhey, 2005). Depression, apathy, and cognitive impairment are very prevalent and significantly contribute to the burden of the disease, but their etiologies remain poorly understood.

The aim of the CASPER study is to gain more insight into the etiologies of post-stroke depression (PSD), post-stroke apathy (PSA), vascular cognitive impairment (VCI), and post-stroke dementia. Therefore, the primary objectives are to identify biomarker-based predictors of PSD, PSA, and VCI. A secondary aim is to study effect modulation, especially the interaction between cerebrovascular disease, neurodegenerative changes and inflammation in post-stroke dementia.

CASPER is a prospective clinical cohort study of 250 first-ever ischemic stroke patients with serial assessments at baseline (10 to 12 weeks after stroke), six and 12 months after baseline. Another wave (36 month after baseline) was later added.

ELIGIBILITY:
Inclusion Criteria:

* First-ever or recurrent ischemic or hemorrhagic stroke
* MMSE score ≥15 (to ensure valid testing)
* Written informed consent
* Sufficient knowledge of the Dutch language
* Preferably participation of an informant

Exclusion Criteria:

* Age younger than 40 years (to exclude atypical strokes)
* Pre-stroke dementia (assessed by a semi-structured interview with a relative, based on clinical diagnosis or IQ-CODE) in the five years prior to stroke
* Psychiatric and neurological disease other than the qualifying event known to affect cognition such as schizophrenia, bipolar disorder, substance abuse, Parkinson's disease, or epilepsy
* Current episode of depression at admission (as evidenced by medical records and patient or informant interview). In contrast, a lifetime history of depression will not be considered as a reason for exclusion as this is considered a potential risk factor for PSD
* Severe aphasia (as it interferes with understanding and following test instructions)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: first-ever and recurrent ischemic and hemorrhagic stroke patients
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
vascular cognitive impairment | 12 months
  defined as a score smaller or equal to 1.5 standard deviations below the general population mean in two or more cognitive domains, based on available norm scores for age, gender and level of education for the Dutch general population
post-stroke depression | 12 months
  measured by the Mini International Neuropsychiatric Interview and the Montgomery-Asberg Depression Rating Scale to assess severity. In addition, the Hospital Anxiety and Depression Scale is used to identify levels of anxiety and depression.
post-stroke apathy | 12 months
  assessed by the Apathy Evaluation Scale (informant- and clinician rated version is used)

SECONDARY OUTCOMES:
change in cognitive function | 12 months
  slope analyses of neuropsychological trajectories in various cognitive domains
incident post-stroke dementia | 12 months
  diagnosed according to the criteria proposed by the National instate of Neurological Disorders and Strokes - Association Internationale pour la Recherch et l'Enseignement en Neurosciences
change in quality of life | 12 months
  measured with the stroke-specific quality of life scale to evaluate health-related quality of life
change in functional ability | 12 months
  measured with the Barthel Index and Lawton questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Köhler, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Netherlands

REFERENCES:
- [Result] Douven E, Schievink SH, Verhey FR, van Oostenbrugge RJ, Aalten P, Staals J, Kohler S. The Cognition and Affect after Stroke - a Prospective Evaluation of Risks (CASPER) study: rationale and design. BMC Neurol. 2016 May 12;16:65. doi: 10.1186/s12883-016-0588-1. PMID 27176617
- [Result] Douven E, Kohler S, Rodriguez MMF, Staals J, Verhey FRJ, Aalten P. Imaging Markers of Post-Stroke Depression and Apathy: a Systematic Review and Meta-Analysis. Neuropsychol Rev. 2017 Sep;27(3):202-219. doi: 10.1007/s11065-017-9356-2. Epub 2017 Aug 22. PMID 28831649
- [Result] Douven E, Kohler S, Schievink SHJ, van Oostenbrugge RJ, Staals J, Verhey FRJ, Aalten P. Temporal Associations between Fatigue, Depression, and Apathy after Stroke: Results of the Cognition and Affect after Stroke, a Prospective Evaluation of Risks Study. Cerebrovasc Dis. 2017;44(5-6):330-337. doi: 10.1159/000481577. Epub 2017 Oct 26. PMID 29073590
- [Result] Douven E, Kohler S, Schievink SHJ, van Oostenbrugge RJ, Staals J, Verhey FRJ, Aalten P. Baseline Vascular Cognitive Impairment Predicts the Course of Apathetic Symptoms After Stroke: The CASPER Study. Am J Geriatr Psychiatry. 2018 Mar;26(3):291-300. doi: 10.1016/j.jagp.2017.09.022. Epub 2017 Sep 28. PMID 29079017
- [Result] Douven E, Aalten P, Staals J, Schievink SHJ, van Oostenbrugge RJ, Verhey FRJ, Kohler S. Co-occurrence of depressive symptoms and executive dysfunction after stroke: associations with brain pathology and prognosis. J Neurol Neurosurg Psychiatry. 2018 Aug;89(8):859-865. doi: 10.1136/jnnp-2017-317548. Epub 2018 Feb 8. PMID 29439160